CLINICAL TRIAL: NCT02925299
Title: An Open-label, Multi-centre, Randomized, Single-period, Parallel Study to Assess the Efficacy, Safety and Utility of 6 Month Day-and-night Automated Closed-loop Insulin Delivery Under Free Living Conditions Compared to Insulin Pump Therapy in Children and Adolescents With Type 1 Diabetes
Brief Title: Day and Night Closed-loop in Young People With Type 1 Diabetes
Acronym: DAN05
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Cambridge University Hospitals NHS Foundation Trust (Other); University of Colorado, Denver (Other); Indiana University (Other); The Leeds Teaching Hospitals NHS Trust (Other); Stanford University (Other); Yale University (Other); Nemours Children's Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAN05; 1UC4DK108520-01 (NIH)
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Endocrine System Diseases; Autoimmune Diseases
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Endocrine System Diseases; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- 24/7 closed loop insulin delivery (Experimental): The study system includes (1) a CGM that measures glucose levels, (2) a computer program on a smartphone that determines how much insulin is needed, and (3) an insulin pump that delivers the insulin. The name of this closed-loop system used in the US is FlorenceM (Medtronic 640G pump and Guardian3 sensor). The name of this closed-loop system in the UK is FlorenceX (DANA pump and Dexcom sensor). Half of the individuals taking part in the study will use the closed-loop study system for 6 months.
  Interventions: Device: FlorenceM (US) and FlorenceX (UK)
- Insulin pump therapy (Active Comparator): Half of the Subjects will continue using their own insulin pump for 6 months.
  Interventions: Device: Insulin pump therapy

INTERVENTIONS:
Device: FlorenceM (US) and FlorenceX (UK) — The automated closed loop system (FlorenceM in US) will consist of:
  Next generation sensor augmented Medtronic insulin pump 640G (Medtronic Minimed, CA, USA) incorporating the Medtronic Guardian3 CGM and glucose suspend feature.
  The automated closed loop system (FlorenceX in UK) will consist of:
  The DANA Diabecare R insulin pump (Sooil Development, Korea) incorporating the Dexcom G6 CGM.
  An Android smartphone containing the Cambridge model predictive algorithm and communicating wirelessly with the insulin pump using a proprietary translator device.
  Arms: 24/7 closed loop insulin delivery
Device: Insulin pump therapy — Subjects will continue using their own insulin pump for 6 months.
  Arms: Insulin pump therapy

SUMMARY:
The main study objective is to determine whether 24/7 automated closed-loop glucose control combined with low glucose feature will improve glucose control as measured by HbA1c.

This is an open-label, multi-centre, multi-national, single-period, randomised, parallel group design study, involving a 6 month period of home study during which day and night glucose levels will be controlled either by a closed-loop system combined with low glucose feature (intervention group) or by insulin pump therapy alone (control group).

It is expected that a total of up to 150 subjects (aiming for 130 randomised subjects) with type 1 diabetes will be recruited through paediatric outpatient diabetes clinics of the investigation centres. Participants will all be on subcutaneous insulin pump therapy.

Subjects in the intervention group will have proven competencies both in the use of the study insulin pump and the study continuous glucose monitoring (CGM) device, and will receive appropriate training in the safe use of closed-loop insulin delivery system and low glucose feature. All subjects will have regular contact with the study team during the home study phase including 24/7 telephone support. The primary outcome is between group differences in HbA1c levels at 6 months post study arm initiation. Secondary outcomes are the time spent in the glucose target (3.9 to 10.0mmol/l; 70 to 180mg/dl), time spent with glucose levels above and below target, as recorded by CGM, and other CGM-based metrics. Safety evaluation comprises assessment of the frequency of severe hypoglycaemic episodes and diabetic ketoacidosis (DKA).

DETAILED DESCRIPTION:
* Purpose of the study: To determine whether 24/7 automated closed-loop glucose control will improve glucose control as measured by glycated haemoglobin and reduce the burden of hypoglycaemia compared to insulin pump therapy alone.
* Study Objectives:

  1. EFFICACY: The objective is to assess efficacy of day and night automated closed-loop glucose control in improving glucose control as measured by glycated haemoglobin, as compared to insulin pump therapy alone.
  2. SAFETY: The objective is to evaluate the safety of day and night automated closed-loop glucose control, in terms of episodes of severe hypoglycaemia and other adverse events.
  3. UTILITY: The objective is to determine the frequency and duration of the use of the automated closed-loop system.
  4. HUMAN FACTORS: The objective is to assess cognitive, emotional, and behavioural characteristics of participating subjects and family members and their response to the closed-loop system and clinical trial using validated surveys and focus groups.
  5. HEALTH ECONOMICS: The objective is to perform a cost utility analysis to inform reimbursement decision-making.
* Study Design: An open-label, multi-centre, randomised, single-period parallel study, contrasting day-and-night automated closed-loop glucose control with insulin pump therapy alone.
* Population: 130 participants randomised (equal proportion of those aged 6 to 12 years and 13 to 18 years, a minimum quota of 25% participants with baseline HbA1c >8.5%)
* Maximum duration of study for a subject: 8 months
* Recruitment: The subjects will be recruited through the pediatric outpatient clinics at each center.
* Consent: Written consent / assent will be obtained from participants and/or guardians according to REC / IRB requirements
* Screening Assessments: Eligible participants will undergo a screening evaluation where blood samples for full blood count, liver, thyroid function and anti-transglutaminase antibodies (with IgA levels if not done within previous 12 months) will be taken. Non-hypoglycaemia C-peptide, glucose and HbA1c will also be measured, and a urine pregnancy test in females of child-bearing potential will be performed.

Surveys investigating participants' quality of life, psychosocial and cognitive functioning, and response to their current treatment will be distributed.

Participants will be fitted with a blinded continuous glucose monitoring (CGM) device to assess baseline glycaemic control. Instructions on how to safely use, remove and send back the device will be provided.

* Study Training: Training sessions on the use of study CGM, insulin pump (and closed loop system for those randomized to be intervention group) will be provided by the research team. Training session on the use of real-time CGM and on how to interpret real-time and retrospective stored data will be provided to all subjects / carers using written material.
* Run-In Period: During a 1-2 week run-in period, subjects will continue using their own insulin pump. Data obtained from blinded CGM and pump downloads may be utilised for therapy adjustment.
* Competency Assessment: Competency on the use of study insulin pump and study CGM will be evaluated using a competency assessment tool developed by the research team. Further training may be delivered as required.
* Randomization: Eligible subjects will be randomised using randomisation software to the use of real-time CGM and low glucose feature combined with day and night closed-loop or to conventional insulin pump therapy alone.

A blood sample will be taken for the measurement of HbA1c and a urine pregnancy test in females of child-bearing potential. A blood sample for centralised analysis of HbA1c will be taken if screening and randomisation are >28 days apart.

1. Automated day and night closed-loop insulin delivery (intervention arm) combined with low glucose feature (interventional arm) - Participants in the closed-loop group will receive additional training sessions following randomisation covering the use of the study insulin pump and real-time CGM, prior to starting closed-loop insulin delivery.

   Once confident with the use of the study pump and CGM system, participants will receive training required for safe and effective use of the closed-loop system approximately 2-4 weeks after randomisation. During this 2-4 hour session participants will operate the system under the supervision of the clinical team. Competency on the use of closed-loop system will be evaluated.

   Thereafter, participants are expected to use closed-loop for 6 months without direct real-time remote monitoring.
2. Insulin pump therapy (control arm) - Refresher training on key aspects of insulin pump therapy will be provided.

Subjects will continue using their own insulin pump for 6 months.

* 3-month and 6 month assessments:

  1. A blood sample will be taken for measurement of HbA1c and a urine pregnancy test in females of child-bearing potential.
  2. Validated surveys evaluating the impact of the devices employed on quality of life, psychosocial and cognitive functioning, diabetes management and treatment satisfaction will be completed.
  3. Participants of both study arms will be fitted with blinded CGM systems at the end of each follow up visit. The sensors will be worn at home for up to 14 days and will be sent back to the research team.

  6 months only: Subjects/guardians will be invited to join follow-up focus groups to gather feedback and reactions to their current treatment (closed-loop or insulin pump), the clinical trial, and quality of life changes.
* Study Contacts: In between study visits, participants will be contacted by the study team (email or phone) once monthly in order to record any adverse events, device deficiencies, and changes in insulin settings, other medical conditions and/or medication.

In case of any technical device or problems related to diabetes management such as hypo- or hyperglycaemia, subjects will be able to contact a 24-hour telephone helpline to the local research team at any time. The local research team will have access to central 24 hour advice on technical issues.

--Procedures for safety monitoring during trial: Standard operating procedures for monitoring and reporting of all adverse events will be in place, including serious adverse events (SAE), serious adverse device effects (SADE) and specific adverse events (AE) such as severe hypoglycaemia.

Subjects will be asked to test and record blood ketones if their finger prick glucose is > 16.7mmol/l (300mg/dl) upon awakening, >300 for more than 1 hour, or >22.2mmo/l (400mg/dL) at any time as part of the safety assessment for DKA.

A data safety and monitoring board (DSMB) will be informed of all serious adverse events and any unanticipated serious adverse device effects that occur during the study and will review compiled adverse event data at periodic intervals.

--Criteria for withdrawal of patients on safety grounds: A subject, parent, or guardian may terminate participation in the study at any time without necessarily giving a reason and without any personal disadvantage. An investigator can stop the closed-loop intervention after consideration of the benefit/risk ratio. Possible reasons are:

1. Serious adverse events
2. Significant protocol violation or non-compliance
3. Failure to satisfy competency assessment
4. Decision by the investigator, or the sponsor, that termination is in the subject's best medical interest
5. Pregnancy, planned pregnancy, or breast feeding
6. Allergic reaction to insulin

Efforts will be made to retain subjects in follow up for the final primary outcome assessment even if the intervention is discontinued, unless the investigator believes that it will be harmful for the subject to continue in the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥6 and <19 years
2. Type 1 diabetes as defined by WHO (51) for at least 1 year [WHO definition: 'The aetiological type named type 1 encompasses the majority of cases with are primarily due to beta-cell destruction, and are prone to ketoacidosis. Type 1 includes those cases attributable to an autoimmune process, as well as those with beta-cell destruction for which neither an aetiology nor a pathogenesis is known (idiopathic). It does not include those forms of beta-cell destruction or failure to which specific causes can be assigned (e.g. cystic fibrosis, mitochondrial defects, etc.).']
3. Use of an insulin pump for at least 3 months, with good knowledge of insulin self-adjustment by subject or caregiver as judged by the investigator
4. Using U-100 rapid acting insulin analogues insulin Aspart or Lispro only
5. Willing to perform regular finger-prick blood glucose monitoring, with at least 4 blood glucose measurements per day day
6. Screening HbA1c ≥ 7.0% (53 mmol/mol) and ≤10 % (86mmol/mol) based on analysis from local laboratory
7. Literate in English
8. Willing to wear glucose sensor
9. Willing to wear closed-loop system at home
10. Willing to follow study specific instructions
11. Willing to upload pump and CGM data at regular intervals
12. Access to WiFi.
13. Lives with someone who is trained to administer intramuscular glucagon and is able to seek emergency assistance

Exclusion Criteria:

1. Living alone
2. Current use of any closed-loop system
3. Any other physical or psychological disease likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator
4. Untreated coeliac disease, adrenal insufficiency, or untreated thyroid disease
5. Current treatment with drugs known to interfere with glucose metabolism, e.g. systemic corticosteroids, non-selective beta-blockers and MAO inhibitors etc.
6. Known or suspected allergy to insulin
7. Clinically significant nephropathy (eGFR < 45ml/min) or on dialysis, neuropathy or active retinopathy (defined as presence of maculopathy or proliferative changes) as judged by the investigator
8. Recurrent incidents of severe hypoglycaemia (>1 episode) during the previous 6 months (adolescents: severe hypoglycaemia is defined as an event requiring assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions including episodes of hypoglycaemia severe enough to cause unconsciousness, seizures or attendance at hospital; children: severe hypoglycaemia is defined as an event associated with a seizure or loss of consciousness)
9. Recurrent incidents of diabetic ketoacidosis (>1 episode) during previous 6 months
10. Unwilling to avoid regular use of acetaminophen
11. Lack of reliable telephone facility for contact
12. Total daily insulin dose ≥ 2 IU/kg/day
13. Total daily insulin dose < 15 IU/day
14. Pregnancy, planned pregnancy, or breast feeding
15. Severe visual impairment
16. Severe hearing impairment
17. Seizure disorder
18. Medically documented allergy towards the adhesive (glue) of plasters or unable to tolerate tape adhesive in the area of sensor placement
19. Serious skin diseases (e.g. psoriasis vulgaris, bacterial skin diseases) located at places of the body, which potentially are possible to be used for localisation of the glucose sensor)
20. Illicit drugs abuse
21. Subject is currently abusing prescription drugs
22. Alcohol abuse
23. Use of pramlintide (Symlin), or other non-insulin glucose lowering agents including sulphonylureas, biguanides, DPP4-Inhibitors, , GLP-1 analogues, SGLT-1/ 2 inhibitors at time of screening
24. Shift work with working hours between 10pm and 8am
25. Sickle cell disease, haemoglobinopathy, or has received red blood cell transfusion or erythropoietin within 3 months prior to time of screening
26. Eating disorder such as anorexia or bulimia
27. Employed by Medtronic Diabetes or with immediate family members employed by Medtronic Diabetes

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 131 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the centralised measurement of glycated haemoglobin (HbA1c) at 6 months. | HbA1c will be taken at baseline, 3 and 6 months
  The objective is to assess efficacy of day and night automated closed-loop glucose control combined with low glucose feature in improving HbA1c, as compared with insulin pump therapy alone.

SECONDARY OUTCOMES:
Time spent in the target glucose range (3.9 to 10mmol/l) (70 to 180mg/dl) | 6 months
  Secondary endpoints regarding glucose levels will be based on sensor glucose data.
Time spent below target glucose (3.9mmol/l)(70mg/dl) | 6 months
  Secondary endpoints regarding glucose levels will be based on sensor glucose data.
Time spent above target glucose (10.0 mmol/l) (180 mg/dl) | 6 months
  Secondary endpoints regarding glucose levels will be based on sensor glucose data.
Mean and standard deviation or percentiles sensor glucose | 6 months
  Secondary endpoints regarding glucose levels will be based on sensor glucose data.
Coefficient of variation of glucose levels | 6 months
  Secondary endpoints regarding glucose levels will be based on sensor glucose data.
Time with glucose levels < 3.5 mmol/l (63 mg/dl) | 6 months
  Secondary endpoints regarding glucose levels will be based on sensor glucose data.
Time with glucose levels <3.0 mmol/l (54 mg/dl) | 6 months
  Secondary endpoints regarding glucose levels will be based on sensor glucose data.
Time with glucose levels in significant hyperglycaemia (glucose levels > 16.7 mmol/l) (300mg/dl) | 6 months
  Secondary endpoints regarding glucose levels will be based on sensor glucose data.
Changes in total basal and bolus insulin dose | 6 months
  Secondary endpoints regarding glucose levels will be based on CRF and insulin pump data.
AUC of glucose below 3.5mmol/l (63mg/dl) | 6 months
  Secondary endpoints regarding glucose levels will be based on sensor glucose data.
AUC glucose above 10.0mmol/L (180mg/dL) | 6 months
  Secondary endpoints regarding glucose levels will be based on sensor glucose data.
HbA1c <7.0%, HbA1c <7.5%, Relative reduction ≥10% from baseline. o Absolute reduction ≥0.5% from baseline o Absolute reduction ≥1% from baseline o Absolute reduction ≥1% from baseline or HbA1c <7.0% | 6 months
  Binary metrics for HbA1c

OTHER OUTCOMES:
Safety Evaluation | 6 months
  Frequency of severe hypoglycaemic episodes as defined by American Diabetes Association (adolescents), and International Society for Pediatric and Adolescent Diabetes (children), frequency of diabetic ketoacidosis (DKA), frequency of severe hyperglycaemia (>16.7 mmol/l)(>300mg/dl) with significant ketosis (plasma ketones >0.6mmol/l) and nature and severity of other adverse events
Utility evaluation | 6 months
  Assessment of the frequency and duration of use of the closed-loop system
Human Factors Assessment | 6 months
  Cognitive, emotional, and behavioural characteristics of participating subjects and family members and their response to the closed-loop system and clinical trial will be assessed gathering both quantitative (validated surveys) and qualitative data (focus groups)
Health Economic Evaluation | 6 months
  Cost utility analysis on the benefits of closed loop insulin delivery to inform reimbursement decision-making

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hovorka, PhD, Study Chair — University of Cambridge; Ajay Thankamony, MD, Principal Investigator — University of Cambridge; Fiona Campbell, MD, Principal Investigator — The Leeds Teaching Hospitals NHS Trust; Bruce Buckingham, MD, Principal Investigator — Stanford University; Stuart Weinzimer, MD, Principal Investigator — Yale University; Linda DiMeglio, MD, Principal Investigator — Indiana University; Paul Wadwa, MD, Principal Investigator — University of Colorado, Denver; Korey Hood, PhD, Principal Investigator — Stanford University; Dana Goldman, PhD, Principal Investigator — University of Southern California; Nikki C Davis, MD, Principal Investigator — Southampton Children's Hospital; Louise Denvir, MD, Principal Investigator — Nottingham Children's Hospital; Nelly Mauras, MD, Principal Investigator — Nemours Children's Health System; Rachel Besser, MD, Principal Investigator — Oxford Children's Hospital; Atrayee Ghatak, MD, Principal Investigator — Alder Hey Children's NHS Foundation Trust
Locations (11):
- United States (5):
  - Stanford University, Palo Alto, California
  - University of Colorado Denver School of Medicine Barbara Davis Center, Aurora, Colorado
  - Yale University, Hartford, Connecticut
  - Nemours Children's Health System, Jacksonville, Florida
  - Indiana University, Indianapolis, Indiana
- United Kingdom (6):
  - University of Cambridge, Cambridge, Cambridgeshire County
  - Nottingham Children's Hospital, Nottingham, England
  - Southampton Children's Hospital, Southampton, England
  - The Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Oxford Children's Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ware J, Boughton CK, Allen JM, Wilinska ME, Tauschmann M, Denvir L, Thankamony A, Campbell FM, Wadwa RP, Buckingham BA, Davis N, DiMeglio LA, Mauras N, Besser REJ, Ghatak A, Weinzimer SA, Hood KK, Fox DS, Kanapka L, Kollman C, Sibayan J, Beck RW, Hovorka R; DAN05 Consortium. Cambridge hybrid closed-loop algorithm in children and adolescents with type 1 diabetes: a multicentre 6-month randomised controlled trial. Lancet Digit Health. 2022 Apr;4(4):e245-e255. doi: 10.1016/S2589-7500(22)00020-6. Epub 2022 Mar 7. PMID 35272971
- [Derived] Musolino G, Allen JM, Hartnell S, Wilinska ME, Tauschmann M, Boughton C, Campbell F, Denvir L, Trevelyan N, Wadwa P, DiMeglio L, Buckingham BA, Weinzimer S, Acerini CL, Hood K, Fox S, Kollman C, Sibayan J, Borgman S, Cheng P, Hovorka R. Assessing the efficacy, safety and utility of 6-month day-and-night automated closed-loop insulin delivery under free-living conditions compared with insulin pump therapy in children and adolescents with type 1 diabetes: an open-label, multicentre, multinational, single-period, randomised, parallel group study protocol. BMJ Open. 2019 Jun 3;9(6):e027856. doi: 10.1136/bmjopen-2018-027856. PMID 31164368